CLINICAL TRIAL: NCT04448782
Title: Characterization of Reverse Triggering and Other Asynchronies in COVID-19 Patients Under Invasive Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Candelaria de Haro, Medical Doctor, Corporacion Parc Tauli
Other Study IDs: RT COVID-19
Record Dates: First submitted 2020-06-17; First posted 2020-06-26 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Asynchronies detection — Asycnhronies detection

SUMMARY:
Prospective observational trial in patients admitted to ICU diagnosed with COVID-19 requiring invasive mechanical ventilation. Characterization of Reverse Triggering asynchrony during the first 5 days of invasive mechanical ventilation and other asynchronies, and its correlation with different outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients under invasive mechanical ventilation more than 24 hours and with a minimum of 48 hours of respiratory signals registered from the ventilator
* Diagnosis of COVID-19

Exclusion Criteria:

* less than 48 hours of data,
* age < 18 years
* admitted from other centers under invasive mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICU under invasive mechanical ventilation with ARDS secondary to COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence and pattern of presentation of Reverse triggering in COVID-19 patients under invasive mechanical ventilation | during the 5 first days of invasive mechanical ventilation
  To analyze the incidence of Reverse Triggering in the initial phases of invasive mechanical ventilation in COVID-19 patients

SECONDARY OUTCOMES:
Incidence of Reverse Triggering related to the level of sedation in COVID-19 patients under invasive mechanical ventilation | From the day of mechanical ventilation initation up to 5 days or the last day of mechanical ventilation
  To correlate the presence of Reverse Triggering with the level of sedation and use of neuromuscular blockers
Reverse triggering and secondary asynchronies in COVID-19 patients under invasive mechanical ventilation | From the day of mechanical ventilation initiation up to 5 days
  To analyze the incidence of breath stacking and ineffective efforts secondary to RT.
Incidence and pattern of presentation of asynchronies in COVID-19 patients under invasive mechanical ventilation | Each day from the day of mechanical ventilation initiation until the day of mechanical ventilation withdrawal or up to 28 days
  To analyze the incidence of RT, ineffective efforts and double triggering throughout the period of invasive mechanical ventilation
Influence of asynchronies in different outcomes in in COVID-19 patients under invasive mechanical ventilation | Each day from the day of mechanical ventilation initiation until the end of invasive mechanical ventilation, ICU discharge and hospital discharge or up to 28 days
  To correlate the presence of asycnhronies and its type with duration of invasive mechanical ventilation, ICU length of stay and survival

CONTACTS AND LOCATIONS:
Locations (1):
- Candelaria de Haro, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided